CLINICAL TRIAL: NCT03820648
Title: Wound Protector Dual-ring Alexis® in Pancreaticoduodenectomy: a Randomized Single-blind Controlled Clinical Trial
Brief Title: Wound Protector Dual-ring Alexis® in Pancreaticoduodenectomy
Acronym: PALEXIS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no differences between the groups at the interim analysis
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE 1369 cesc
Record Dates: First submitted 2018-09-26; First posted 2019-01-29 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2019-12

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: The study is an RCT, single-blinded, conducts in patients with cancer submitted to PD (1:1). In the experimental group, we will use the dual-ring WP Alexis (Applied Medical, Rancho Santa Margarita, California, USA), while in the control group we will use the standard 3M™ Steri-Drape 2. There is planned a clinical visit of follow-up on the 30th day from the operation day (as in clinical practice).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alexis® device (Experimental): In this group, we will be used WP dual-ring Alexis® (Figure 1). The Alexis® 's size will be decided on the basis of abdominal incision (Alexis® X-Large or Alexis® XX-Large will be used for 11-17cm or 17-25 cm incision length respectively)
  Interventions: Device: Alexis
- Standard 3M™ Steri-Drape 2 (Active Comparator): In this group, we will be used Standard 3M™ Steri-Drape 2
  Interventions: Device: Standard 3M™ Steri-Drape 2

INTERVENTIONS:
Device: Alexis — The Alexis® (Applied Medical) is a surgical device indicated for use in retracting and protecting an incision during laparoscopic or open surgery. It is intended to allow the surgeon to access through an atraumatic circumferentially 360 degrees retracted wound that provides maximum exposure with minimum incision size. Further, once positioned, the Alexis Wound Retractor is intended to protect against wound contamination.The device will be manufactured in five sizes, extra-small, small, medium, medium-large and large. The Alexis Wound Retractor has been found non-toxic and non-irritant when tested in accordance with ISO 10993, Part 1: Biological Evaluation of Medical Devices. The materials used in the manufacturing of the Alexis Wound Retractor have been tested in accordance with applicable standards and was determined to pass tensile strength, elongation, (ASTM D 412) and Tear Strength (ASTM D 624). Functional performance testing has been completed and has passed the required testing.
  Arms: Alexis® device
Device: Standard 3M™ Steri-Drape 2 — Standard 3M™ Steri-Drape 2 is a standard drape applicated on the skin of the patient before the surgical incision.
  Arms: Standard 3M™ Steri-Drape 2

SUMMARY:
Surgical site infection (SSI) is a leading cause of preventable morbidity and mortality in North America and worldwide. This condition has consistently been reported to account for up to 25% of all healthcare-associated infections. In a cost analysis, SSIs post-pancreaticoduodenectomy (PD) dramatically increases the treatment costs. More importantly, postoperative wound infections delay postoperative adjuvant chemotherapy, which is indicated in the majority of patients undergoing PD for pancreatic cancer. Protective covers or 'wound protectors' are hypothesized to be an improvement over adhesive membrane barriers as they are believed to reduce intraoperative contamination while concomitantly preserving the temperature and humidity of the surgical wound. The aim of this study is to assess if the use of wound protector can reduce the wound infection rate in patients undergoing to PD.

DETAILED DESCRIPTION:
Surgical site infection (SSI) is a leading cause of preventable morbidity and mortality in North America and worldwide. This condition has consistently been reported to account for up to 25% of all healthcare-associated infections. Prolonged hospitalization, more frequent hospital re-admissions after surgery and a greater than twofold increase in costs and mortality have consistently been associated with this condition over the past decade. The SSI is associated with an increased risk of postsurgical pain, poor wound healing and aesthetic results and an increased risk of incisional hernias. The literature shows an incidence rate of SSI at 30 days after surgery that reaches 51% of cases. In particular, the incidence of wound infection is 15%. In our experience, the rate of wound infection in patients undergoing Pancreaticoduodenectomy (PD) is 10%.

SSI is an infectious process that is localized to surgical incision level and it is classified as being either incisional or organ/space. Incisional SSI is further divided into those involving only skin and subcutaneous tissue (superficial incisional SSI) and those involving deeper soft tissues of the incision (deep incisional SSI).

In a cost analysis, SSIs post-PD dramatically increases the treatment costs. More importantly, postoperative wound infections delay postoperative adjuvant chemotherapy, which is indicated in the majority of patients undergoing PD for pancreatic cancer. During recent years there is also an increasing incidence of antibiotic-resistant pathogens in hospitals, so several studies have suggested primary or secondary prevention strategies to reduce SSI rate. In order to minimize the risk of SSI, various measures of perioperative care have already been adopted, including the cleaning of the skin, the hair removal of the intervention area, the prevention of intraoperative hypothermia and perioperative antibiotic therapy. However there are few studies on the effectiveness of surgical procedures for primary prevention to reduce the contamination in the surgical site, especially in patients undergoing major gastrointestinal surgery. The surgical procedures classified as contaminated or dirty (with a higher bacterial load within the surgical site and/or regarding gastrointestinal or biliary tracts) remain associated with an increased risk of SSI, about two times, compared to the interventions classified as clean or clean-contaminated. The PD is classified as surgery contaminated / dirty.

The use of adhesive membrane barriers over the skin of the surgical site emerged 50 years ago as a possible solution to minimize endogenous cross-contamination during surgery. The initial idea relied on the principle of reducing exposure of the surgical site to bacteria inherent in the surrounding skin or to airborne bacteria in the operating room. Major applicability was expected in clean surgeries, where the skin is considered the main source of bacteria. Unfortunately, however, no evidence in support of plastic adhesive drapes was found in a recently updated systematic review of randomized controlled trials (RCTs) including five studies and 3082 patients. In fact, a 23% increase in the risk of SSI was found in the group that received adhesive drapes. In the 1960s, other devices were described and then developed based on the concept of combining a non-traumatic surgical wound retractor with a protective membrane covering of the incisional margin in abdominal surgeries. Such protective covers or 'wound protectors' (WP) were hypothesized to be an improvement over adhesive membrane barriers as they were believed to reduce intraoperative contamination while concomitantly preserving the temperature and humidity of the surgical wound. In support of this hypothesis, early studies demonstrated reduced exposure of the surgical wound to enteric bacteria at the end of gastrointestinal operations. These results were further supported by several RCTs, which demonstrated that wound protectors were efficacious in reducing the incidence of incisional SSI as compared to usual care in patients undergoing gastrointestinal surgeries. A recently meta-analysis of RCTs on the WP enrolled 6 studies and 1008 patients, finding that the pooled estimated risk of SSI among patients fitted with wound protectors during surgery was 0.55 (95% CI 0.31 to 0.98) times the pooled estimated risk of SSI in control groups.

The aim of this study is to assess if the use of WP can reduce the wound infection rate in patients undergoing to PD.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective PD
* Age ≥ 18 years
* Ability of the subject to understand character and individual consequences of the clinical trial
* Written informed consent

Exclusion Criteria:

* Under 18 years of age
* Unable to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | 30th day postoperative
  Number of SSI onset in patients submitted to PD until the 30th day postoperative. This endpoint will be compared between the two groups.

SECONDARY OUTCOMES:
Device resistance | Intraoperative
  Number intraoperative device rupture in both groups. It will be also recorded the number of device lesions seen at the end of the surgical operation.
Treatment costs related to increased hospital stays due to SSI | 30th day postoperative
  Number of additional days to the average hospital stays (7 days) of the patients submitted to PD at our Institute, related to the onset of SSI until the 30th day postoperative
Costs related to the use of additional antibiotics administered for the treatment of SSI | 30th day postoperative
  Evaluation of the total costs of the additional antibiotic therapy administered for the treatment of SSI, developed within the 30th day postoperative, in the two patient groups. It will be considered like the ex-factory price of the drug.

CONTACTS AND LOCATIONS:
Locations (1):
- AOUI Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Pastena M, Marchegiani G, Paiella S, Fontana M, Esposito A, Casetti L, Secchettin E, Manzini G, Bassi C, Salvia R. Use of an intraoperative wound protector to prevent surgical-site infection after pancreatoduodenectomy: randomized clinical trial. Br J Surg. 2020 Aug;107(9):1107-1113. doi: 10.1002/bjs.11527. Epub 2020 Mar 12. PMID 32162321